CLINICAL TRIAL: NCT05337280
Title: Feasibility of Assessing Breast Cancer Neoadjuvant Therapy Response Using Imagio Opto-Acoustic Imaging
Brief Title: OA for Breast Cancer NAC Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seno Medical Instruments Inc. (Industry)
Collaborators: American College of Radiology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Device Feasibility
Other Study IDs: NEO-01
Record Dates: First submitted 2022-02-10; First posted 2022-04-20 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a single center sequential design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Imagio OA/US (Experimental): Imagio OA/US Imaging
  Interventions: Device: Imagio OA/US

INTERVENTIONS:
Device: Imagio OA/US — Imagio optoacoustic/ultrasound

SUMMARY:
This is an early research and development study. The objective of this study is to determine the feasibility of the Imagio OA/US Breast Imaging System to detect complete breast cancer pathologic response to neoadjuvant therapy as assessed by functional optoacoustic features, vascular features and relative degrees of oxygenation/deoxygenation

DETAILED DESCRIPTION:
The use of neoadjuvant systemic therapy in the treatment of breast cancer patients is increasing beyond the scope of locally advanced disease. Imaging provides important information in assessing response to therapy as a complement to conventional tumor measurements via physical examination. Tumor response to neoadjuvant therapy can also provide prognostic information. As stated in the background section, the attainment of pCR after completion of neoadjuvant therapy and surgical resection is associated with improved disease-free survival [1-3]. This correlation is especially strong for Triple-receptor negative (ER, PR negative and HER-2 non amplified), and HER-2 positive breast cancer. Studies of neoadjuvant therapy have used a variety of methods for assessing tumor response. Currently, there are no established clinical practice guidelines for how best to assess tumor response to neoadjuvant therapy. Typically, patients undergo conventional breast imaging (mammography and US) and physical examination, and DCE-MRI in selected cases.

The Imagio OA/US technology is an alternative imaging technology that demonstrates both gray scale ultrasound morphologic information, including size measurements, and functional information that includes presence or absence of tumor angiogenesis, degree of angiogenesis, and relative degrees of oxygenation and deoxygenation of hemoglobin.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years and older male or female patients;
2. Ipsilateral intact biopsy-proven invasive breast cancer clinical T1-T4 (by standard of care imaging), including primary or recurrent disease.
3. Patient eligible to receive neoadjuvant chemotherapy

Exclusion Criteria:

1. Known Stage IV disease (breast or other cancer);
2. Have a condition or impediment (i.e., insect bites, poison ivy, open sores, chafing of the skin, scar, tattoos, moles, etc.); that could interfere with the intended field of view (within one probe length or 4 cm of the nodule);
3. Patient has received chemotherapy for any type of cancer within 90 days from date of baseline Imagio OA/US exam;
4. Is experiencing photo-toxicity associated with currently taking, or having taken, photosensitizing agents within the previous 72 hours such as sulfa, ampicillin, tetracycline;
5. Is currently undergoing phototherapy;
6. Has a history of any photosensitive disease (e.g., porphyria, lupus erythematosus);
7. Is undergoing treatment for a photosensitive disease and is experiencing photosensitivity;
8. Pregnancy;
9. Patient has participated in a clinical study of an investigational drug or device within 3 months prior to screening visit that may have an impact on clinical outcomes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2023-01-04 (Actual)

PRIMARY OUTCOMES:
The number of masses that may exhibit qualitative changes in accordance with Functional Feature Scale as assessed by Imagio OA/US over the course of baseline though follow-up timepoints | Baseline to Post Surgical Assessment at 6 months
  Feature scores per mass derived per Feature Score Scale (0-6 and 0-5 scoring- lower score mean most likely benign) per 5 mass features (External Peripheral Zone, External Capsular Boundary, Internal Shape, Internal Echotexture, Internal Sound ) used to predict number of masses that demonstrated response or no response at all time points (baseline, cycle 2, mid cycle and pre surgical) to chemotherapy treatment
Number of masses that correlate with chemotherapy response/no response as assessed by Functional Feature Score Scale at all study timepoints to predict optimal timing for Imagio imaging | Baseline to Post Surgical Assessment at 6 months
  Number of masses assessed at baseline and follow-up timepoints - cycle 2, mid cycle and pre surgical f/u that correlate with feature score (External Peripheral Zone, External Capsular, Internal Vessel Score, Internal Total Hemoglobin, Internal Deoxygenated Blush) changes assessed by Feature Score Scale (0-6 nd 0-5 scores depending on feature) and pathologic complete response (pCR) to determine optimal timing for imaging.

OTHER OUTCOMES:
Number of metastatic lymph nodes scored using a Lymph Node Scoring Scale that may correlate with chemotherapy response | Baseline to Post Surgical Assessment at 6 months
  Imagio OA/US imaging of metastatic lymph nodes will be assessed using a designated Lymph Node Scale (Shape Score, Cortical Thickness, Margin Score and Hilar Compression Score, Size Score) to predict response(0 = benign / 1 = benign, uncertain / 2-4 = probably malignant / >=5 = malignant) to chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Basak Dogan, MD, Principal Investigator — UT Southwestern
Locations (1):
- UT Southwestern, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No